CLINICAL TRIAL: NCT07275021
Title: The Vision Study: Cerebral/ Cortical Visual Impairment (CVI)
Brief Title: Cerebral/ Cortical Visual Impairment: Screening, Identification and Outcome Prediction in Neonates
Acronym: CVI
Status: Recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Mohamed El-Dib, MD, Director, Neonatal Neurocritical Care Department of Pediatrics, Division of Newborn Medicine, Brigham and Women's Hospital Associate Professor of Pediatrics, Harvard Medical School President, Newborn Brain Society, Brigham and Women's Hospital
Other Study IDs: 2025P001413
Record Dates: First submitted 2025-08-19; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-08

CONDITIONS: Preterm Less Than 32wks With IVH, WMI/PVL; Late Preterm or Term (37-42wks) With Neonatal Encephalopathy Treated With Hypothermia for HIE
Keywords: Cerebral/ Cortical Visual Impairment; Vision Disorders, Cerebral/Cortical; Brain Injuries; Visual Disorders; Periventricular Leukomalacia; Hypoxic-Ischemic Encephalopathy; Hypoxia-Ischemia, Brain; White Matter Injury; Visual Evoked Potentials; Infant, Extremely Premature (for <32 weeks GA); Germinal Matrix Hemorrhage; Intraventricular Hemorrhage; Neonatal Encephalopathy; Prenatal Stroke
MeSH Terms: conditions — Vision Disorders; Brain Injuries; Leukomalacia, Periventricular; Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preterm/Term High-Risk Infants: Infants at high risk for Cerebral/Cortical Visual Impairment (CVI), including preterm infants with IVH or white matter injury, term or late preterm infants with hypoxic-ischemic encephalopathy (HIE), and infants with perinatal stroke. Participants are followed prospectively and undergo standardized clinical, neuroimaging, neurophysiologic, and developmental assessments through 24 months of age.
  Interventions: Other: Prospective Clinical and Neurodevelopmental Data Collection

INTERVENTIONS:
Other: Prospective Clinical and Neurodevelopmental Data Collection — Participants undergo standardized collection of clinical, neuroimaging, neurophysiologic, visual assessment and neurodevelopmental data as part of this prospective observational study. Data include information obtained from clinical care and scheduled follow-up assessments through 24 months of age. No interventions are assigned.

SUMMARY:
Cerebral/Cortical Visual Impairment (CVI) is the leading cause of childhood visual impairment in the United States and other industrialized countries. CVI is a brain-based visual disorder in which visual acuity or visual fields are reduced despite a normal eye examination or greater-than-expected visual impairment relative to ocular pathology. CVI is increasingly recognized in children with neurological conditions, yet it often remains undiagnosed until later childhood, delaying opportunities for early intervention.

Population-based studies suggest that CVI is more common than previously understood. Recent estimates indicate that over 180,000 individuals in the United States aged 0-22 years may have diagnosed or likely CVI, with only a minority formally identified. Children with CVI frequently have co-occurring neurological conditions, including cerebral palsy, epilepsy, developmental delays, or genetic disorders. Infants born preterm or with conditions such as hypoxic-ischemic encephalopathy (HIE), perinatal stroke, or white matter injury are at particularly high risk. Prospective research also shows that a substantial proportion of infants born very preterm exhibit behavioral features of CVI later in childhood.

Despite improvements in neonatal neurocritical care, early detection of CVI remains challenging. Current clinical practice focuses on managing conditions such as HIE, perinatal stroke, periventricular leukomalacia, and other brain injuries, but there is limited research evaluating structured early identification pathways for CVI in infancy. Diagnostic tools such as brain MRI and Visual Evoked Potentials (VEP) have shown potential for identifying brain-based visual dysfunction, but their integration into early predictive models for CVI has not been fully explored.

This study addresses a critical gap in pediatric care by prospectively evaluating high-risk neonates using clinical, neuroimaging, neurophysiologic, and standardized developmental assessments through 24 months of age. Early identification of CVI may support timely referral for visual rehabilitation and developmental services, potentially improving long-term functional outcomes. Developing a predictive model for early CVI detection will contribute to improved clinical pathways, enhance early diagnosis, and reduce the long-term educational and social burden associated with undetected CVI. Ultimately, this research aims to improve outcomes and quality of life for infants at risk for brain-based visual impairment.

DETAILED DESCRIPTION:
The study is a prospective observational study designed to follow preterm and term infants who are at high risk for Cerebral/ Cortical Visual Impairment (CVI). Preterm Infants born before 32 weeks gestational age with conditions such germinal matrix/intraventricular hemorrhage (IVH), white matter injury (WMI including periventricular leukomalacia (PVL), and late term and term infants with Hypoxic-Ischemic Encephalopathy (HIE) or prenatal Stroke will be enrolled during the neonatal intensive care unit (NICU) stay and monitored through a structured follow-up schedule. The study focuses on data collection using advanced diagnostic imaging and neurodevelopmental assessments without introducing randomization or experimental interventions.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born < 32 weeks gestational age with any of the following:
* Germinal matrix/intraventricular hemorrhage (IVH)
* White matter injury (WMI), including periventricular leukomalacia (PVL)
* Late preterm infants (born 34-36 weeks gestation) or term infants (born 37-42 weeks gestation) with:
* Neonatal encephalopathy treated with therapeutic hypothermia for suspected hypoxic-ischemic encephalopathy (HIE)
* Infants diagnosed with perinatal stroke

Parent(s) or legal guardian(s) willing and able to provide informed consent

Exclusion Criteria:

Neonates whose parent(s) or guardian(s) cannot commit to long-term follow-up

Ages: 31 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — All genders are eligible to participate.
Study Population: The study population includes preterm and term infants at high risk for cerebral visual impairment due to neurological injury diagnosed in the neonatal period. This includes:
  * Preterm infants born <32 weeks gestation with intraventricular hemorrhage or white matter injury
  * Late preterm (34-36 weeks) and term (37-42 weeks) infants with hypoxic-ischemic encephalopathy treated with therapeutic hypothermia or diagnosed with perinatal stroke
  Eligible infants are enrolled during their initial hospitalization and followed longitudinally into early childhood to assess visual development, neurodevelopmental outcomes, and early signs of cerebral visual impairment. Parent(s) or legal guardian(s) must be willing and able to provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of Cerebral Visual Impairment (CVI) at 24 Months | 24 months of age
  Diagnosis of Cerebral/Cortical Visual Impairment (CVI) based on standardized clinical visual assessment performed.
  Outcome measure: Low, or high risk.

SECONDARY OUTCOMES:
Visual Function assessment | 24 months
  Visual function evaluated using the age-appropriate CVI and parent questionnaire administered at scheduled follow-up intervals (6, 12, and 24 months per protocol), with primary reporting at 24 months.
  * Teller acuity Cards (testing distance: 38 cms, 55 cms 84 cms)
  * Patti Pics or grating acuity (testing distance: 25 cms, 50 cms and 100 cms)
  * Visual behavior scale (grade: 1, 2, or 3)
  * Resolution Distance Visual acuity
  Outcome measure: Low, or high risk.
Visual Evoked Potential (VEP) Response | 24 months
  Assessment of cortical visual pathway response using VEP performed at 6 and 24 months per protocol, with primary reporting at 24 months. Outcome measure: low or high risk group.
Neurodevelopmental Composite Score | 24 months
  Standardized neurodevelopmental testing obtained as part of 12-, 18-, and 24-month clinical follow-up (e.g., Bayley-IV). Primary reporting at 24 months
  Outcome measure:
  * Low-Risk: scores within or above age-expected norms
  * High-Risk: scores ≥1 SD below the mean (Standard Score <85) indicating developmental delay

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed El-Dib, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, and Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data

REFERENCES:
- [Background] Chang MY, Borchert MS. Advances in the evaluation and management of cortical/cerebral visual impairment in children. Surv Ophthalmol. 2020 Nov-Dec;65(6):708-724. doi: 10.1016/j.survophthal.2020.03.001. Epub 2020 Mar 19. PMID 32199940
- [Background] Pilling RF, Allen L, Bowman R, Ravenscroft J, Saunders KJ, Williams C. Clinical assessment, investigation, diagnosis and initial management of cerebral visual impairment: a consensus practice guide. Eye (Lond). 2023 Jul;37(10):1958-1965. doi: 10.1038/s41433-022-02261-6. Epub 2022 Oct 18. PMID 36258009
- [Background] Sakki HEA, Dale NJ, Sargent J, Perez-Roche T, Bowman R. Is there consensus in defining childhood cerebral visual impairment? A systematic review of terminology and definitions. Br J Ophthalmol. 2018 Apr;102(4):424-432. doi: 10.1136/bjophthalmol-2017-310694. Epub 2017 Nov 16. PMID 29146757